CLINICAL TRIAL: NCT05818410
Title: Human-Prosthetic Interaction: Brain & Technology After Lower-Limb Loss
Acronym: HumanIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Kevin De Pauw, Prof. Dr., Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EC-2023-089
Record Dates: First submitted 2022-12-14; First posted 2023-04-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries | interventions — Artificial Limbs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- New prosthesis (Experimental): 20 participants will be fitted with the Lunaris foot and follow the protocol
  Interventions: Device: Prosthetic device (Lunaris)
- Standard prosthesis (Active Comparator): 20 participants will be fitted with the SACH foot and follow the protocol
  Interventions: Device: Prosthetic device (Sach foot)
- Control group of able-bodied individuals (Other): 20 able-bodied individuals will be recruited to enable comparison with both groups of participants with lower limb amputation
  Interventions: Other: No prosthetic device

INTERVENTIONS:
Device: Prosthetic device (Lunaris) — Participants with an amputation will conduct experiments with the prosthetic device
  Arms: New prosthesis
Other: No prosthetic device — Able-bodied individuals will conduct experiments to enable comparison with the participants with amputation
  Arms: Control group of able-bodied individuals
Device: Prosthetic device (Sach foot) — Participants with an amputation will conduct experiments with the prosthetic device
  Arms: Standard prosthesis

SUMMARY:
This study evaluates brain neuroplasticity and functional performance in people with unilateral lower limb amputation.

DETAILED DESCRIPTION:
The researchers will investigate the beneficial effect of a passive prosthetic ankle (Lunaris®) on functional physical performance, brain neuroplasticity and movement patterns compared to conventional prosthetic feet and able-bodied individuals.

The clinical trial will comprise four test days for participants with a lower limb amputation and two days for the control group of able-bodied individuals.

The able-bodied individuals will undergo an MRI scan at the University Hospital Brussels (dpt. Radiology and Magnetic Resonance) and perform functional performance tests.

Participants with a lower limb amputation will start the clinical trial upon the start of their rehabilitation. At week 0, when initiating the rehabilitation, participants will undergo a baseline MRI scan at the University Hospital Brussels (dpt. Radiology and Magnetic Resonance). Then, they will be allocated to the intervention arms (Lunaris® or the SACH foot®) and will conduct their rehabilitation to learn to walk with a prosthesis. At the end of the rehabilitation, after 12 weeks, participants will perform baseline functional performance tests, fill out the prosthetic evaluation questionnaire (PEQ) measuring the quality of life. Between weeks 12 and 24 of the clinical trial (i.e. intervention period), participants will perform their daily activities with the allocated prosthesis. During weeks 12 - 24, trying out new prosthetic devices will be allowed within the group of individuals wearing the SACH foot® as this is considered the usual care. At the end of this period (after week 24), the post-test assessment will take place and participants will undergo the same MRI and functional performance tests and fill out the PEQ as during the baseline assessments to evaluate the changes that occurred. Additionally, participants will be asked to fill out the Quebec User Evaluation of Satisfaction with Assistive Technology. The 12-week intervention period is chosen based on a study examining the effect of 12 weeks of balance training in healthy and older adults on neuroplasticity and the accommodation time to walking with a new prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial (below knee) amputation
* Healthy subject
* Medicare Functional Classification Level: K3-4

Exclusion Criteria:

* Any neurological disease
* Upper limb or bilateral amputation
* Osso-integration
* Metal implants
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Brain neuroplasticity | Change over 24 weeks
  Brain scan: diffusion-weighted imaging

SECONDARY OUTCOMES:
Performance | Change over 12 weeks
  time (seconds) to complete L-test
Performance | Change over 12 weeks
  time (seconds) to complete dual-L test
Performance | Change over 12 weeks
  time (seconds) to complete slope walking test
Performance | Change over 12 weeks
  time (seconds) to complete stair climbing test
Performance | Change over 12 weeks
  Accuracy of the dual-L-test in percent
Biomechanical | Change over 12 weeks
  Continious relative phase thigh [calculated from the hip & knee joint angles and velocities]
Biomechanical | Change over 12 weeks
  Continious relative phase knee-ankle calculated from the knee-ankle joint angles and velocities (Lamb et al, 2014)
Performance | Change over 12 weeks
  Distance covered during the 6-minute walk test
Psychological | Change over 12 weeks
  Score on the prosthetic evaluation questionnaire
Psychological | Change over 12 weeks
  Visual analogue scale for comfort (score: 0= not comfortable, 100 = comfortable) and fatigue (score: 0= not fatiguing, 100 = fatiguing) during all tasks
Psychological | Change over 12 weeks
  Borg rating of perceived exertion (score: 6 = No exertion at all , 20 = Maximal exertion)
Psychological | Change over 12 weeks
  Perceived workload: Nasa-Task Load Index (score: 0 = minimal workload, 100 = Maximal perceived workload )

CONTACTS AND LOCATIONS:
Overall Officials: Kevin De Pauw, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox PD, Frengopoulos CA, Hunter SW, Sealy CM, Deathe AB, Payne MWC. Impact of Course Configuration on 6-Minute Walk Test Performance of People with Lower Extremity Amputations. Physiother Can. 2017;69(3):197-203. doi: 10.3138/ptc.2016-24. PMID 30275635
- [Background] Howard CL, Wallace C, Perry B, Stokic DS. Comparison of mobility and user satisfaction between a microprocessor knee and a standard prosthetic knee: a summary of seven single-subject trials. Int J Rehabil Res. 2018 Mar;41(1):63-73. doi: 10.1097/MRR.0000000000000267. PMID 29293160
- [Background] Windrich M, Grimmer M, Christ O, Rinderknecht S, Beckerle P. Active lower limb prosthetics: a systematic review of design issues and solutions. Biomed Eng Online. 2016 Dec 19;15(Suppl 3):140. doi: 10.1186/s12938-016-0284-9. PMID 28105948
- [Background] Russell Esposito E, Aldridge Whitehead JM, Wilken JM. Step-to-step transition work during level and inclined walking using passive and powered ankle-foot prostheses. Prosthet Orthot Int. 2016 Jun;40(3):311-9. doi: 10.1177/0309364614564021. Epub 2015 Jan 27. PMID 25628378
- [Background] Molina-Rueda F, Navarro-Fernandez C, Cuesta-Gomez A, Alguacil-Diego IM, Molero-Sanchez A, Carratala-Tejada M. Neuroplasticity Modifications Following a Lower-Limb Amputation: A Systematic Review. PM R. 2019 Dec;11(12):1326-1334. doi: 10.1002/pmrj.12167. Epub 2019 Jun 18. PMID 30989836
- [Background] Boone DA, Coleman KL. Use of the Prosthesis Evaluation Questionnaire (PEQ). JPO: Journal of Prosthetics and Orthotics. 2006;18(6).
- [Background] Ozer S, Young J, Champ C, Burke M. A systematic review of the diagnostic test accuracy of brief cognitive tests to detect amnestic mild cognitive impairment. Int J Geriatr Psychiatry. 2016 Nov;31(11):1139-1150. doi: 10.1002/gps.4444. Epub 2016 Feb 18. PMID 26891238
- [Background] Rogge AK, Roder B, Zech A, Hotting K. Exercise-induced neuroplasticity: Balance training increases cortical thickness in visual and vestibular cortical regions. Neuroimage. 2018 Oct 1;179:471-479. doi: 10.1016/j.neuroimage.2018.06.065. Epub 2018 Jun 26. PMID 29959048
- [Background] Rogge AK, Roder B, Zech A, Nagel V, Hollander K, Braumann KM, Hotting K. Balance training improves memory and spatial cognition in healthy adults. Sci Rep. 2017 Jul 18;7(1):5661. doi: 10.1038/s41598-017-06071-9. PMID 28720898
- [Background] Mahon CE, Hendershot BD. Biomechanical accommodation to walking with an ankle-foot prosthesis: An exploratory analysis of novice users with transtibial limb loss within the first year of ambulation. Prosthet Orthot Int. 2022 Oct 1;46(5):452-458. doi: 10.1097/PXR.0000000000000124. Epub 2022 Mar 25. PMID 35333820
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Hart SG, Staveland LE. Development of NASA-TLX (Task Load Index): Results of Empirical and Theoretical Research. In: Hancock PA, Meshkati N, editors. Advances in Psychology. 52: North-Holland; 1988. p. 139-83.
- [Background] Agrawal V, Gailey RS, Gaunaurd IA, O'Toole C, Finnieston A, Tolchin R. Comparison of four different categories of prosthetic feet during ramp ambulation in unilateral transtibial amputees. Prosthet Orthot Int. 2015 Oct;39(5):380-9. doi: 10.1177/0309364614536762. Epub 2014 Jun 12. PMID 24925671
- [Background] Schmalz T, Blumentritt S, Marx B. Biomechanical analysis of stair ambulation in lower limb amputees. Gait Posture. 2007 Feb;25(2):267-78. doi: 10.1016/j.gaitpost.2006.04.008. Epub 2006 May 24. PMID 16725325
- [Background] Hunter SW, Frengopoulos C, Holmes J, Viana R, Payne MW. Determining Reliability of a Dual-Task Functional Mobility Protocol for Individuals With Lower Extremity Amputation. Arch Phys Med Rehabil. 2018 Apr;99(4):707-712. doi: 10.1016/j.apmr.2017.12.008. Epub 2018 Jan 6. PMID 29317224
- [Background] Cho YS, Jang SH, Cho JS, Kim MJ, Lee HD, Lee SY, Moon SB. Evaluation of Validity and Reliability of Inertial Measurement Unit-Based Gait Analysis Systems. Ann Rehabil Med. 2018 Dec;42(6):872-883. doi: 10.5535/arm.2018.42.6.872. Epub 2018 Dec 28. PMID 30613081
- [Background] Kong XZ, Liu Z, Huang L, Wang X, Yang Z, Zhou G, Zhen Z, Liu J. Mapping Individual Brain Networks Using Statistical Similarity in Regional Morphology from MRI. PLoS One. 2015 Nov 4;10(11):e0141840. doi: 10.1371/journal.pone.0141840. eCollection 2015. PMID 26536598
- [Background] Tzourio-Mazoyer N, Landeau B, Papathanassiou D, Crivello F, Etard O, Delcroix N, Mazoyer B, Joliot M. Automated anatomical labeling of activations in SPM using a macroscopic anatomical parcellation of the MNI MRI single-subject brain. Neuroimage. 2002 Jan;15(1):273-89. doi: 10.1006/nimg.2001.0978. PMID 11771995
- [Background] Peterson SM, Ferris DP. Group-level cortical and muscular connectivity during perturbations to walking and standing balance. Neuroimage. 2019 Sep;198:93-103. doi: 10.1016/j.neuroimage.2019.05.038. Epub 2019 May 18. PMID 31112786
- [Background] Lamb PF, Stockl M. On the use of continuous relative phase: Review of current approaches and outline for a new standard. Clin Biomech (Bristol). 2014 May;29(5):484-93. doi: 10.1016/j.clinbiomech.2014.03.008. Epub 2014 Mar 26. PMID 24726779
- [Background] Aledda S, Galeoto G, Fabbrini G, Lucibello L, Tofani M, Conte A, Berardi A. A systematic review of the psychometric properties of Quebec user evaluation of satisfaction with assistive technology (QUEST). Disabil Rehabil Assist Technol. 2024 May;19(4):1228-1235. doi: 10.1080/17483107.2022.2161648. Epub 2023 Jan 16. PMID 36645802
- [Derived] Lathouwers E, Tassignon B, Maricot A, Radwan A, Naeyaert M, Raeymaekers H, Van Schuerbeek P, Sunaert S, De Mey J, De Pauw K. Human-Prosthetic Interaction (HumanIT): A study protocol for a clinical trial evaluating brain neuroplasticity and functional performance after lower limb loss. PLoS One. 2024 Mar 21;19(3):e0299869. doi: 10.1371/journal.pone.0299869. eCollection 2024. PMID 38512879